CLINICAL TRIAL: NCT04238910
Title: Maximizing Energy After Traumatic Brain Injury: Feasibility and Effectiveness of Combined Problem Solving Therapy and Occupational Therapist Delivered Education
Brief Title: Maximizing Energy After Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ketki Raina, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO09010275; W81XWH-10-1-0 (Other Grant/Funding Number: US Army Medical Research and Development Command)
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2020-01

CONDITIONS: Traumatic Brain Injury; Fatigue
Keywords: traumatic brain injury; fatigue; self-management
MeSH Terms: conditions — Brain Injuries, Traumatic; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maximizing Energy (Experimental): The Maximizing Energy (MAX) intervention consists of two weekly 30-minute sessions delivered live via the Internet using web-camera technology for 8 weeks. The interventions are delivered by occupational therapists.
  The MAX intervention was developed by combining two active ingredients - Problem Solving Therapy and energy conservation strategy education. Participants engage in two introductory sessions during the first week of the intervention. During the first session in a week, participants practice the steps of MAX Intervention with a fatigue-related problem. At the end of the session, the participants identify a clearly defined action plan for solution implementation. Participants are asked to implement the solution over the next few days. The second session takes place later in the week. The interventionist reviews the problem, the identified solution, and its implementation. Participants use a workbook to support their application of the MAX Intervention.
  Interventions: Behavioral: Maximizing Energy
- Health Education (Active Comparator): consists of two weekly 30-minute sessions delivered live via the Internet using web-camera technology for 8 weeks. The interventionist delivered health education using a variety of health related topics relevant to individuals with TBI (e.g., characteristics and prevalence of fatigue after TBI, diet and nutrition, importance of exercise, energy conservation strategies).Participants use a workbook to follow along with the interventionist during the weekly sessions.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Maximizing Energy — The intent of the MAX intervention is to personalize OT delivered education to facilitate the implementation of Energy Conservation strategies using the PST framework to address specific fatigue-related problems and then to generalize from these solutions to both similar and new situations in daily life.
  Arms: Maximizing Energy
Behavioral: Health Education — The intent of the health education intervention is to control for the non-specific effects of interactions with an interventionist. Participants received education on a variety of health related topics relevant to individuals with TBI.
  Arms: Health Education

SUMMARY:
Traumatic brain injury (TBI) is the signature injury of the wars in Iraq and Afghanistan. Up to 73% of TBI patients endorse fatigue as their most challenging symptom.

Fatigue leads to decreased participation in everyday life and return to work. The Maximizing Energy (MAX) intervention trains individuals with TBI to manage their fatigue.

The intervention individualizes the Occupational Therapist delivered Energy Conservation Strategies education by using the framework of Problem Solving Therapy. The purpose of this single-blind randomized clinical trial was to test the effect of the Maximizing Energy (MAX) intervention for decreasing the impact and severity of post-TBI fatigue, increasing participation in everyday life and physical activity, and decreasing work disability.

DETAILED DESCRIPTION:
A significant proportion (50-80%) of individuals with traumatic brain injury (TBI) experience persistent fatigue and endorse it as the most distressing and challenging symptom that affects daily life. Chronic fatigue has a devastating impact on individuals because it leads to reduced participation in everyday life. Despite the high incidence of post-TBI fatigue and its impact on everyday life, these is a dearth of studies examining the effectiveness of non-pharmacological interventions for the treatment of post-TBI fatigue. This study is unique in that it will examine the effectiveness of a non-pharmacological intervention to manage post-TBI fatigue. The Maximizing Energy (MAX) Intervention, individuals with post-TBI fatigue will reduce the impact of fatigue on everyday life by actively seeking and implementing solutions for their fatigue-related problems, thus promoting their reintegration into the community.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years or older
2. Patient lives within a 50 miles radius of the University of Pittsburgh in Oakland
3. Diagnosis of TBI atleast 6 months ago: Individuals need time to determine if they have chronic fatigue after CA.
4. Community dwelling: Community dwelling participants are more likely to be able to make environmental changes than those in institutions
5. Vision to operate a computer:
6. Presence of fatigue: Fatigue Severity Scale is a valid and reliable test used to measure the severity of fatigue on 9 fatigue-related statements on a 7 point ordinal scale. A score ≥ 4 signifies fatigue severe enough to limit daily activities.
7. No cognitive impairment
8. Functional English fluency and literacy

Exclusion Criteria:

1. Physical impairment: Individuals scoring < 65 on the 13 Functional Independence Measure (FIM) motor items will be excluded from the study;
2. Mood and mental health history: Individuals with a recent (less than 3 months) history of major depressive disorder, mania, hypomania, psychosis, or substance abuse as diagnosed by the PRIME-MD and the MiniInternational Neuropsychiatric Interview (MINI) unless treated or in partial remission will be excluded because their self-reports of participation in everyday life may not be reliable; and
3. Disability due to other diagnoses: history of neurologic, traumatic, or psychiatric conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue Scores (Patient-Reported Outcomes Measurement Information System - Fatigue) Between Groups At 16 Weeks | Baseline, Week 16
  The PROMIS Fatigue item banks assess a range of self-reported fatigue symptoms that likely decreases one's ability to execute daily activities and function normally in family or social roles. The computerized adaptive test version provides a mean fatigue score. The Scale uses a T-score metric in which 50 is the mean for the population and 10 is the standard deviation of that population. Higher scores equal more fatigue. Scores were obtained at baseline, Week 8, Week 12, and Week 16 for each participant, and mean scores were calculated for each group at each time point.

SECONDARY OUTCOMES:
Change in Fatigue Impact Scores (Modified Fatigue Impact Scale) Between Groups At 16 Weeks | Baseline, Week 16
  The Modified Fatigue Impact Scale is a self-report instrument that assesses the impact of fatigue on performance of everyday activities. The Scale has 21 items in three subscales: physical, cognitive, and psychosocial. A 5-point scale ranging from 0 (never) to 4 (almost always) is used for rating each item; items are summed to obtain a total score. Higher scores indicate greater impact of fatigue on performance of everyday activities. Total scores were obtained at baseline, Week 8, Week 12, and Week 16 for each participant, and mean scores were calculated for each group at each time point.
Change in Fatigue Severity Scores (Fatigue Severity Scale) Between Groups At 16 Weeks | Baseline, Week 16
  The Modified Fatigue Severity Scale is a self-report instrument that assesses the severity of fatigue. The Scale has 9 items. A 7-point scale ranging from 1 (strong disagreement) to 7 (strong agreement) is used for rating each item; mean of the items yield a total score. Higher scores indicate greater fatigue severity. Total scores were obtained at baseline, Week 8, Week 12, and Week 16 for each participant, and mean scores were calculated for each group at each time point.
Change in Participation Scores (Participation Objective, Participation Subjective) Between Groups At 16 Weeks | Baseline, Week 16
  Participation Objective, Participation Subjective (POPS) evaluates participation in everyday life in persons with TBI. The scale consists of 26 items sorted into five categories: Domestic life; Major life activities; Transportation; Interpersonal interactions and relationships; and Community, recreational and civic life. Scores on the objective questions are converted into standardized z scores ranging from -3 to +3. Higher scores indicate greater frequency of participation in everyday life. Scores on the subjective questions range from +4, indicating a "most important" area of life that the person is engaging in at a satisfactory level, to -4, indicating an equally important area of life that the person wants to do either less of or more of. Total scores were obtained at baseline, Week 8, Week 12, and Week 16 for each participant, and mean scores were calculated for each group at each time point.
Change in Physical Activity Between Groups At 16 Weeks | Baseline, Week 16
  Physical activity data was collected with the Actical device. The Actical is a wireless, wearable body monitor that collects and analyzes raw physiological and lifestyle data. It was worn at the wrist for 3 days. Physical activity data was derived in terms of metabolic equivalents (METs) when participants engaged in physical activity. Total energy expenditure over 3 days were obtained at at baseline, Week 8, Week 12, and Week 16 for each participant, and mean scores were calculated for each group at each time point.
Change in Perceived Work Disability (Work Role Functioning Questionnaire) Between Groups At 16 Weeks | Baseline, Week 16
  The Work Role Functioning Questionnaire (WRFQ) assesses the degree of perceived work disability due to a chronic health problem. The questionnaire consists of 27 items divided into five subscales: Work scheduling demands, Physical demands, Mental demands, Social demands, and Output demands. The participant scores each item on a 5 point ordinal scale (0 = difficult all the time, 4 = difficult none of the time). Each subscale is scored separately, by adding the response of each item, and converting the score from 0 (limited all the time) to 100 (never limited).

CONTACTS AND LOCATIONS:
Overall Officials: Ketki Raina, PhD, OTR/L, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raina KD, Morse JQ, Chisholm D, Leibold ML, Shen J, Whyte E. Feasibility of a Cognitive Behavioral Intervention to Manage Fatigue in Individuals With Traumatic Brain Injury: A Pilot Study. J Head Trauma Rehabil. 2016 Sep-Oct;31(5):E41-9. doi: 10.1097/HTR.0000000000000196. PMID 26580691